CLINICAL TRIAL: NCT01185938
Title: Protective Effect of Rosuvastatin and Antiplatelet Therapy On Contrast-induced Nephropathy and Myocardial Damage in Patients With Acute Coronary Syndrome Undergoing Coronary Intervention; PRATO-ACS Trial
Brief Title: Statin Contrast Induced Nephropathy Prevention
Acronym: PRATO-ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiopatici Toscani (Other)
Responsible Party: Principal Investigator, Anna Toso, MD, Centro Cardiopatici Toscani
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 552010
Record Dates: First submitted 2010-08-03; First posted 2010-08-20 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Acute Coronary Syndrome
Keywords: statin; CIN; periprocedural damage
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Control (No Intervention)

INTERVENTIONS:
Drug: Rosuvastatin — One oral single dose of rosuvastatin of 40 mg at admission and then 20 mg/day for 1 month.
  Arms: Rosuvastatin

SUMMARY:
This open-label study, prospective, randomized trial evaluating the acute (in-hospital) pleiotropic and clinical effects of a hydrophilic statin (rosuvastatin) in patients with acute coronary syndrome

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether, in patients with acute coronary syndromes not taking statins in chronic administration, high doses of a hydrophilic statin (rosuvastatin) administered before coronary angiography and/or angioplasty, may exert a renal-protective effect by reducing the incidence of contrast nephropathy. Contrast induced nephropathy is defined as increased values of creatinine >= 0.3 mg/dl from baseline values, within 72 hours after contrast medium exposure.

Secondary end points: 1) verify if short-term (<48 hours)statin administration reduces the peak levels and the curve areas of markers of myocardial necrosis throughout the hospitalization period and if reduces the occurrence of periprocedural infarction. Biochemical markers (quantitative creatine kinase-MB (CK-MB) mass and Troponin I) are measured at admission and at 6, 12, and 24 hours during the first day then once daily, immediately before angiography, and 24 hours thereafter. In patients who underwent coronary angioplasty (PCI), biochemical markers were measured at 12 and 24 hours after the procedure. Data were fitted, peak values and curve areas calculated; the occurrence of periprocedural infarction was defined as a CK-MB mass elevation more than three times the upper limit of normal within 24 hours after PCI. 2) determine the distribution of peripheral lymphocytic populations at the entry and at discharge using the flow cytometric analysis; 3) analyze the clinical composite outcome of death, myocardial infarction, urgent revascularization, dialysis and stroke at 30 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Are eligible for the study all patients admitted to CCU for Acute Coronary Syndrome without ST elevation (NSTEMI) candidates for early invasive strategy (coronary angiography within 48 hours from the admission) and without previous therapy with statins.

Exclusion Criteria:

1. inability to provide consent
2. pregnancy or lactation
3. intolerance to statins
4. therapy with other lipid lowering drugs
5. acute or chronic liver disease
6. chronic muscle disease
7. acute renal failure or chronic renal failure stage IV
8. neoplastic
9. exposure to iodinated contrast medium in the previous 10 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy in patients with Acute Coronary Syndrome treated with rosuvastatin versus control | 3 days

SECONDARY OUTCOMES:
Peak levels and curve areas of myocardial necrosis markers measured throughout the hospitalization period. | 5 days (average)
  Quantitative creatine kinase-MB (CK-MB) mass and cTn I were measured at admission and at 6, 12, and 24 hours during the first day then once daily, immediately before angiography, and 24 hours thereafter. In patients who underwent angioplasty, biochemical markers were measured at 12 and 24 hours after procedure.
Distribution of peripheral lymphocyte populations at the entry and at discharge | 5 days (average)
  Comparison between groups for the distribution of peripheral lymphocyte sub-population evaluated bu Flow Cytometric Analysis at the admission and at discharge.
Incidence of clinical composite outcome (death, myocardial infarction, urgent revascularization, dialysis and stroke). | 30 days and 6 months
  Clinical follow-up at 30 days and 6 month after the hospitalization for the Acute Coronary Syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Toso, MD, Study Chair — Misericordia e Dolce, Prato Hospital, Cardiology Unit
Locations (1):
- Cardiology Division, Prato Hospital, Prato, Prato, Italy

REFERENCES:
- [Derived] Toso A, Leoncini M, Maioli M, Tropeano F, Di Vincenzo E, Villani S, Bellandi F. Relationship between inflammation and benefits of early high-dose rosuvastatin on contrast-induced nephropathy in patients with acute coronary syndrome: the pathophysiological link in the PRATO-ACS study (Protective Effect of Rosuvastatin and Antiplatelet Therapy on Contrast-Induced Nephropathy and Myocardial Damage in Patients With Acute Coronary Syndrome Undergoing Coronary Intervention). JACC Cardiovasc Interv. 2014 Dec;7(12):1421-9. doi: 10.1016/j.jcin.2014.06.023. PMID 25523533
- [Derived] Leoncini M, Toso A, Maioli M, Tropeano F, Badia T, Villani S, Bellandi F. Early high-dose rosuvastatin and cardioprotection in the protective effect of rosuvastatin and antiplatelet therapy on contrast-induced acute kidney injury and myocardial damage in patients with acute coronary syndrome (PRATO-ACS) study. Am Heart J. 2014 Nov;168(5):792-7. doi: 10.1016/j.ahj.2014.08.005. Epub 2014 Aug 10. PMID 25440809
- [Derived] Leoncini M, Toso A, Maioli M, Tropeano F, Villani S, Bellandi F. Early high-dose rosuvastatin for contrast-induced nephropathy prevention in acute coronary syndrome: Results from the PRATO-ACS Study (Protective Effect of Rosuvastatin and Antiplatelet Therapy On contrast-induced acute kidney injury and myocardial damage in patients with Acute Coronary Syndrome). J Am Coll Cardiol. 2014 Jan 7-14;63(1):71-9. doi: 10.1016/j.jacc.2013.04.105. Epub 2013 Sep 26. PMID 24076283